CLINICAL TRIAL: NCT00407849
Title: Phase I/II Study of Intravitreal Triamcinolone Acetonide Microspheres for Treatment of Diffuse Diabetic Macular Edema Unresponsive to Conventional Laser Photocoagulation Treatment.
Brief Title: Intravitreal Triamcinolone Acetonide for Treatment of Refractory Diffuse Diabetic Macular Edema
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Federal University of Sao Paulo, Vision Institute Department of Ophthalmology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RETAAC001
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: triamcinolone acetonide — Intravitreal injection

SUMMARY:
Phase I/II study with intravitreal triamcinolone acetonide microspheres(RETAAC)for treatment of diffuse diabetic macular edema unresponsive to laser photocoagulation. Study hypothesis is that single intravitreal injection of RETAAC is safe and efficient compared to conventional treatment. Fifty patients will participate in this study and will be randomized into treatment and observation groups. Efficacy will be evaluated by best corrected visual acuity and macular thickness measured by optic coherence tomography (OCT) after 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or 2)
* Diabetic macular edema in study eye associated to diabetic retinopathy
* Diffuse macular edema defined as macular thickening determined by biomicroscopy and fluorescein angiography.
* Best corrected visual acuity between 34 (20/200) and 68 letters (20/50).
* Macular thickness greater than 300 mcm on OCT.

Exclusion Criteria:

* Uncontrolled systemic disease
* Start of medical therapy for diabetes or change in treatment from oral to insulin four months before initial visit.
* HbA1c levels greater than 10%
* Presence of retinal venous occlusion, cystoid macular edema,or other condition that would contribute to macular edema.
* Presence of epiretinal membrane
* Presence of vitreomacular traction in the study eye.
* Aphakic or anterior chamber intraocular lens in the study eye.
* Neovascularization of disc or elsewhere in the study eye.
* History or presence of choroidal neovascularization in the study eye.
* Presence of rubeosis irides in the study eye.
* Eye opacity that interfere with clinical documentation and photography.
* Intra-ocular surgery 90 days before initial visit.
* Previous vitrectomy in study eye.
* Previous history of intravitreal or periocular corticoid or any other intravitreal drug in study eye.
* Scheduled surgery for study eye.
* Patients with known allergies to fluorescein, iodo-povidone or any component of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity after 12 months of single intravitreal injection of triamcinolone acetonide. | 12 months
Macular thickness measured by optical coherence tomography (OCT) after 12 months of treatment. | 12 months
Safety of intravitreal triamcinolone acetonide after 12 months of treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Cardillo, M.D, Principal Investigator — Federal University of São Paulo
Locations (1):
- Vision Institute, Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Martidis A, Duker JS, Greenberg PB, Rogers AH, Puliafito CA, Reichel E, Baumal C. Intravitreal triamcinolone for refractory diabetic macular edema. Ophthalmology. 2002 May;109(5):920-7. doi: 10.1016/s0161-6420(02)00975-2. PMID 11986098
- [Background] Massin P, Audren F, Haouchine B, Erginay A, Bergmann JF, Benosman R, Caulin C, Gaudric A. Intravitreal triamcinolone acetonide for diabetic diffuse macular edema: preliminary results of a prospective controlled trial. Ophthalmology. 2004 Feb;111(2):218-24; discussion 224-5. doi: 10.1016/j.ophtha.2003.05.037. PMID 15019365
- [Background] Gillies MC, Sutter FK, Simpson JM, Larsson J, Ali H, Zhu M. Intravitreal triamcinolone for refractory diabetic macular edema: two-year results of a double-masked, placebo-controlled, randomized clinical trial. Ophthalmology. 2006 Sep;113(9):1533-8. doi: 10.1016/j.ophtha.2006.02.065. Epub 2006 Jul 7. PMID 16828501